CLINICAL TRIAL: NCT00497666
Title: Retrospective Study Evaluating the Association Between Rosiglitazone Use and Clinical Course of Diabetic Nephropathy: Population-Based Study
Brief Title: Association Between Rosiglitazone Use and Clinical Course of Diabetic Nephropathy: Population-Based Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 346147Rosi
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-07

CONDITIONS: Diabetes; Diabetic Nephropathy; Renal Protection
Keywords: Diabetes; Diabetic nephropathy; renal protection
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitasone (retrospective observation)

SUMMARY:
Recent data show that Rosiglitazone treatment can reduce proteinuria in diabetic patients. However, currently there are no trials that examine the effects of Rosiglitazone on kidney disease progression, that is, doubling of serum creatinine or time to onset of end-stage renal disease, in patients with diabetic nephropathy.

We decided to study retrospectively the possible association between rosiglitazone use and clinical course of diabetic nephropathy, including rate of deterioration of renal function, appearance and progression of microalbuminuria/proteinuria, survival and acceptance to renal replacement therapy.

DETAILED DESCRIPTION:
Background Type 2 diabetes mellitus is a public health concern, and projections of its future effect are alarming. According to the World Health Organization, diabetes affects more than 170 million people worldwide, and this number will rise to 370 million by 2030 [1]. About one third of those affected will eventually have progressive deterioration of renal function [2, 3]. The first clinical sign of renal dysfunction in patients with diabetes is generally microalbuminuria (a sign of endothelial dysfunction that is not necessarily confined to the kidney)[4], which develops in 2 to 5 percent of patients per year [5,6]. In type 2 diabetes, unlike type 1 diabetes [7], microalbuminuria is seldom reversible [8], but, instead, progresses to overt proteinuria in 20 to 40 percent of patients.[9,10]. In 10 to 50 percent of patients with proteinuria, chronic kidney disease develops that ultimately requires dialysis or transplantation [11,12,13]. Forty to 50 percent of patients with type 2 diabetes who have microalbuminuria eventually die of cardiovascular disease [14,15]; this is three times as high a rate of death from cardiac causes as among patients who have diabetes but have no evidence of renal disease [6].

In patients with diabetes and renal disease, lowering blood pressure and the levels of urinary albumin is effective in reducing the risk of end-stage renal disease as well as that of myocardial infarction, heart failure, and stroke [16]. Angiotensin-converting-enzyme (ACE) inhibitors or angiotensin II antagonists appear to be the most effective renoprotective and antihypertensive agents [11, 12, 17-21] . Treatment with the ACE inhibitor enalapril over a period of six years decreased the incidence of microalbuminuria in patients with type 2 diabetes who were normotensive and not obese [22].

Preventing (or delaying) the development of microalbuminuria is a key treatment goal for renoprotection [23] and, possibly, for cardioprotection [4]. Recent clinical trials suggested that inhibition of the renin-angiotensin system may actually prevent nephropathy. The post hoc analyses of the reduction in hypertension in the Heart Outcomes Prevention Evaluation study [18] and in the Losartan Intervention for Endpoint study [24] found a lower incidence of overt nephropathy in subjects with type 2 diabetes who received therapy that inhibited the renin-angiotensin system than in controls.

Recent BENEDICT study indicates that treatment with trandolapril with or without verapamil significantly reduces the incidence of microalbuminuria in patients with type 2 diabetes and normal urinary albumin excretion, as compared with placebo [25]. Trandolapril alone also appeared to decrease the incidence of microalbuminuria, whereas verapamil had no effect. Thiseffect of trandolapril plus verapamil and trandolapril alone in preventing microalbuminuria exceeded expectations based on changes in blood pressure alone.

Unfortunately, even with the appropriate use of available therapy, diabetic nephropathy still remains the leading cause of ESRD [2]. More effective strategies are needed in order to retard the progression of diabetic nephropathy and to reduce cardiovascular mortality in diabetic population.

Thiazolidinediones (TZDs) represent a class of compounds currently used for the treatment of type 2 DM that exert their hypoglycemic properties through reduction of IR [26]. These agents act by stimulating a certain type of nuclear receptor, called peroxisome proliferator-activated receptor gamma (PPAR ). Such receptors are abundant in adipose tissue cells, but they are also present in various other cell types, such as vascular smooth muscle cells, macrophages, vascular endothelial cells, colon epithelial cells, as well as renal glomerular and tubular cells. Through transcriptional regulation of various genes, PPAR receptors play an important role in adipocyte differentiation and lipid and carbohydrate metabolism [26]. Apart from improving glycemic control in patients with type 2 DM, several lines of evidence support the notion that TZDs have beneficial effects on other components of the metabolic syndrome, such as blood pressure (BP) lowering, triglyceride reduction, high-density lipoprotein-cholesterol elevation, redistribution of body fat away from the central compartment, decrease of C-reactive protein and plasminogen activator inhibitor -1 (PAI-1) levels, and others [26].

Additionally, several animal studies demonstrate that TZDs also reduce urine albumin or protein excretion and protect against injury to the kidney [27]. Moreover, experimental studies exposed numerous actions of TZDs in the kidney that could explain a possible renoprotective effect [27-30]. Our recent study on diabetic rats showed that rosiglitazone exerts its anti-inflammatory renoprotective effect by inhibition of mesangial cells proliferation, downregulation of apoptosis and blunting responsiveness to angiotensin-2 [31].

Human study also report significant reductions in UAE among patients with type 2 diabetes by rosiglitazone [32].

Another human study was part of a cardiac safety study where rosiglitazone 4 mg b.i.d. was compared to glyburide in 121 patients for 52 weeks [32]. After 28 weeks of treatment, both groups had significant reductions in ACR of about 30%, but after 52 weeks only rosiglitazone group continued to demonstrate a significant ACR reduction. This finding suggests that duration of follow-up is an important variable in assessing the effect of TZDs [32].

Overall, the above data clearly show that TZD treatment can reduce UAE. However, it should be emphasized that currently there are no trials that examine the effects of TZDs on kidney disease progression, that is, doubling of serum creatinine or time to onset of end-stage renal disease, in patients with diabetic nephropathy [33]. Such studies are needed in order to provide the best evidence for a renoprotective effect of TZDs.

Based on this data, we decided to study the possible association between rosiglitazone use and clinical course of diabetic nephropathy, including rate of deterioration of renal function, appearance and progression of microalbuminuria/proteinuria, survival and acceptance to renal replacement therapy.

Methods. Study population. The study is planned as retrospective cohort study using automated clinical data of Central Region Clalit Health Survices from 1999 until 2007.

Inclusion criteria: 1. Diagnosis of Diabetes Mellitus Type II; 2. Treatment With Oral hypoglycemics; 3. Availability of Baseline and follow up clinical data Exclusion criteria: 1. Insulin Therapy at baseline; 2. Malignancy Patients will be divided into 2 groups: rosiglitazone-treated group and non-treated with rosiglitazone ( control) group.

Baseline Data ( separately for two groups). Number of patients. Gender Race/etnicity Age Weight, BMI Duration of DM Diabetic microangiopathy: retinopathy, neuropathy, nephropathy Medications for DM Creatinine Microalbumin Proteinuria HbA1c% Hb Ca, P, PTH Albumin Hypertension: BP Cholesterol, LDL, TG Smoking: current, previous Alcohol consumption Comorbidites: HTN, CAD, CHF, PVD, Hypercholesterolemia, CVA/TIA Drugs: ACEi, ARBs, CCB, beta-blockers, statines, antiplatlate Use of nephrotoxic medications: NSAIDs

Follow up data Duration of rosiglitasone therapy/follow up Use of contrast media during study

Every year data:

Creatinine eGFR Microalbumin Proteinuria HbA1C% Start of insulin therapy

Events:

Hospitalisation (cause) Death (cause) ESRD/Dialysis Reported CHF MI CVA Angiography PVD Amputation References

1. World Health Organization. The Diabetes Program 2004. (at http://www.who.int/diabetes/en/.)
2. Remuzzi G, Schieppati A, Ruggenenti P. Nephropathy in patients with type 2 diabetes. N Engl J Med 2002;346:1145-1151.
3. Ruggenenti P, Remuzzi G. The diagnosis of renal involvement in non-insulin-dependent diabetes mellitus. Curr Opin Nephrol Hypertens 1997;6:141-145.
4. Ritz E. Albuminuria and vascular damage -- the vicious twins. N Engl J Med 2003;348:2349-2352.
5. Gall MA, Hougaard P, Borch-Johnsen K, Parving HH. Risk factors for development of incipient and overt diabetic nephropathy in patients with non-insulin dependent diabetes mellitus: prospective, observational study. BMJ 1997;314:783-788.
6. Adler AI, Stevens RJ, Manley SE, Bilous RW, Cull CA, Holman RR. Development and progression of nephropathy in type 2 diabetes: the United Kingdom Prospective Diabetes Study (UKPDS 64). Kidney Int 2003;63:225-232.
7. Perkins BA, Ficociello LH, Silva KH, Finkelstein DM, Warram JH, Krolewski AS. Regression of microalbuminuria in type 1 diabetes. N Engl J Med 2003;348:2285-2293
8. Parving HH, Lehnert H, Brochner-Mortensen J, Gomis R, Andersen S, Arner P. The effect of irbesartan on the development of diabetic nephropathy in patients with type 2 diabetes. N Engl J Med 2001;345:870-878
9. Mogensen CE. Microalbuminuria predicts clinical proteinuria and early mortality in maturity-onset diabetes. N Engl J Med 1984;310:356-360
10. Nelson RG, Knowler WC, Pettitt DJ, Saad MF, Charles MA, Bennett PH. Assessing risk of overt nephropathy in diabetic patients from albumin excretion in untimed urine specimens. Arch Intern Med 1991;151:1761-1765.
11. Brenner BM, Cooper ME, de Zeeuw D, et al. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. N Engl J Med 2001;345:861-869.
12. Lewis EJ, Hunsicker LG, Clarke WR, et al. Renoprotective effect of the angiotensin receptor antagonist irbesartan in patients with nephropathy due to type 2 diabetes. N Engl J Med 2001;345:851-860.
13. Nelson RG, Newman JM, Knowler WC, et al. Incidence of end-stage renal disease in type 2 (non-insulin-dependent) diabetes mellitus in Pima Indians. Diabetologia 1988;31:730-736
14. Eurich DT, Majumdar SR, Tsuyuki RT, Johnson JA. Reduced mortality associated with the use of ACE inhibitors in patients with type 2 diabetes. Diabetes Care 2004;27:1330-1334.
15. Parving HH, Mauer M, Ritz E. Diabetic nephropathy. In: Brenner BM, ed. Brenner & Rector's The kidney. 7th ed. Vol. 2. Philadelphia: Saunders, 2004:1777-818.
16. Dinneen SF, Gerstein HC. The association of microalbuminuria and mortality in non-insulin-dependent diabetes mellitus: a systematic overview of the literature. Arch Intern Med 1997;157:1413-1418
17. Parving HH, Jacobsen P, Rossing K, Smidt UM, Hommel E, Rossing P. Benefits of long-term antihypertensive treatment on prognosis in diabetic nephropathy. Kidney Int 1996;49:1778-1782
18. Heart Outcomes Prevention Evaluation (HOPE) Study Investigators. Effects of ramipril on cardiovascular and microvascular outcomes in people with diabetes melllitus: results of the HOPE study and MICRO-HOPE substudy. Lancet 2000;355:253-259. [Erratum, Lancet 2000;356:860.]
19. Viberti G, Mogensen CE, Groop LC, Pauls JF. Effect of captopril on progression to clinical proteinuria in patients with insulin-dependent diabetes mellitus and microalbuminuria. JAMA 1994;271:275-279.
20. Ravid M, Lang R, Rachmani R, Lishner M. Long-term renoprotective effect of angiotensin-converting enzyme inhibition in non-insulin-dependent diabetes mellitus: a 7-year follow-up study. Arch Intern Med 1996;156:286-289
21. Lewis EJ, Hunsicker LG, Bain RF, Rohde RD. The effect of angiotensin-converting-enzyme inhibition on diabetic nephropathy. N Engl J Med 1993;329:1456-1462. [Erratum, N Engl J Med 1993;330:152.
22. Ravid M, Brosh D, Levi Z, Bar-Dayan Y, Ravid D, Rachmani R. Use of enalapril to attenuate decline in renal function in normotensive, normoalbuminuric patients with type 2 diabetes mellitus: a randomized, controlled trial. Ann Intern Med 1998;128:982-988
23. UK Prospective Diabetes Study (UKPDS) Group. Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). Lancet 1998;352:837-853. [Erratum, Lancet 1999;354:602.]
24. Lindholm LH, Ibsen H, Dahlof B, et al. Cardiovascular morbidity and mortality in patients with diabetes in the Losartan Intervention For Endpoint reduction in hypertension study (LIFE): a randomized trial against atenolol. Lancet 2002;359:1004-1010.
25. Ruggenenti P, Fassi A, Ilieva A, et al. Preventing Microalbuminuria in Type 2 Diabetes. N Engl J Med 2004; 351: 1941-51.
26. Lebovitz HE, Banerji MA. Insulin resistance and its treatment by thiazolidinediones. Recent Prog Horm Res 2001; 56: 265-294.
27. Haneda M, Koya D, Kikkawa R. Cellular mechanisms in the development and progression of diabetic nephropathy: activation of the DAG-PKC-ERK pathway. Am J Kidney Dis 2001; 38: S178-S181
28. Asano T, Wakisaka M, Yoshinari M et al. Peroxisome proliferator-activated receptor gamma1 (PPARgamma1) expresses in rat mesangial cells and PPARgamma agonists modulate its differentiation. Biochim Biophys Acta 2000; 1497: 148-154
29. Xiong Z, Huang H, Li J et al. Anti-inflammatory effect of PPARgamma in cultured human mesangial cells. Renal Failure 2004; 26: 497-505.
30. Gumieniczek A. Effect of the new thiazolidinedione-pioglitazone on the development of oxidative stress in liver and kidney of diabetic rabbits. Life Sci 2003; 74: 553-562
31. Weissgarten J, Berman S, Efrati S, et al. Apoptosis and proliferation of cultured mesangial cell isolated from kidneys of rosiglitasone-treated pregnant diabetic rats. Nephrol Dial Transplant 2006; 21: 1198-204
32. Bakris G, Viberti G, Weston WM et al. Rosiglitazone reduces urinary albumin excretion in type 2 diabetes. J Hum Hypertens 2003; 17: 7-12.
33. Sarafidis P, Bakris G. Protection of the kidney by thiazolidinediones: An assessment from bench to bedside. Kidney Int 2006; 70: 1223-1233.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Diabetes Mellitus Type II
2. Treatment With Oral hypoglycemics
3. Availability of Baseline and follow up clinical data

Exclusion Criteria:

1. Insulin Therapy at baseline
2. Malignancy

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-08; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Leonid S Feldman, Principal Investigator — Nephrology Division, Assaf Harofeh Medical Center, Zerifin,; Leonid S Feldman, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Clalit Health Cervices, Central District, Ẕerifin, Israel